CLINICAL TRIAL: NCT05798117
Title: An Open-label, Multi-center, Phase 1/2 Study to Assess Safety, Efficacy and Cellular Kinetics of YTB323 in Participants With Severe, Refractory Systemic Lupus Erythematosus
Brief Title: An Open-label, Study to Assess Safety, Efficacy and Cellular Kinetics of YTB323 in Severe, Refractory Systemic Lupus Erythematosus
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYTB323G12101; 2022-001796-14 (EudraCT Number)
Record Dates: First submitted 2023-02-27; First posted 2023-04-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
Keywords: CAR-T, YTB323, Lupus, SLE, LN, severe refractory SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- YTB323 (Experimental): Single infusion of YTB323
  Interventions: Drug: YTB323

INTERVENTIONS:
Drug: YTB323 — Single infusion of YTB323

SUMMARY:
The study is intended to assess safety, efficacy and cellular kinetics of YTB323 treatment in participants with severe refractory systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adequate renal, hepatic, cardiac, hematological and pulmonary function
* Men and women with SLE, aged ≥18 years and ≤65 years at screening, fulfilling the 2019 European League Against Rheumatism EULAR/ACR classification criteria for SLE.
* Patient must be positive for at least one of the following autoantibodies at screening: antinuclear antibodies (ANA) at a titer of ≥1:80, or anti dsDNA (above the ULN); or anti-Sm (above the ULN)
* Active (severe) disease as defined by SLEDAI-2K ≥ 8 (not including the SLEDAI-2K domains of lupus headache, cerebrovascular accident, organic brain syndrome) and at least one of the following significant SLE related organ involvements:
* Renal
* At least moderate or severe peri/myocarditis
* At least moderate or severe pleuritis or other lung involvement
* Vasculitis
* Failure to respond to two or more standard immunosuppressive therapies (including one of mycophenolate or cyclophosphamide), unless contraindicated or having experienced documented adverse events or intolerance related to such immunosuppressive drugs not allowing their further use, in combination with glucocorticoids and failure to respond to at least one biological agent (unless contraindicated, the patient deemed ineligible by the Investigator or not available in a country).

Exclusion Criteria:

* Clinically significant active, opportunistic, chronic or recurrent infection confirmed by clinical evidence, imaging, or positive laboratory tests (e.g., blood cultures, PCR for DNA/RNA, such as COVID-19 etc.) one month prior to or during screening. Patients who have had at least one severe infection that required prolonged hospitalization in the intensive care setting within 5 years prior to screening and/or at least one severe infection that required prolonged hospitalization within one year prior to screening.
* Uncontrolled diabetes mellitus, lung diseases or any other illness that are not related to SLE that in the opinion of the Investigator would jeopardize the ability of the patient to tolerate lymphodepletion and CD19 CAR-T cell therapy
* Prior history of malignancy except for localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis
* Any patients requiring medications prohibited by the protocol
* Any psychiatric condition or disability making compliance with treatment or informed consent impossible
* Prior treatment with anti-CD19 therapy, adoptive T cell therapy or any prior gene therapy product (e.g. CAR-T cell therapy)
* History of bone marrow/hematopoietic stem cell or solid organ transplantation
* Female participants who are pregnant or breastfeeding, or intending to conceive during the course of the study
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using a highly effective method of contraception starting from the time of enrollment to at least 12 months after the YTB323 infusion (or longer if required as per local regulations) and until CAR-T cells are no longer present by qPCR on two consecutive tests
* Sexually active males unwilling to use a condom during intercourse from the time enrollment for at least 12 months after the YTB323 infusion and until CAR-T cells are no longer present by qPCR on two consecutive tests
* Any acute, severe lupus related flare during screening that needs immediate treatment and/or makes the immunosuppressive washout impossible; thus, makes the patient ineligible for CD19 CAR-T therapy as judged by the Investigator, such as acute central nervous system (CNS) lupus (e.g. psychosis, epilepsy) or catastrophic antiphospholipid syndrome
* Significant, likely irreversible organ damage related to SLE, e.g. end stage renal disease, that in the opinion of the Investigator renders CD19 CAR-T cell therapy would be unlikely to benefit the patient
* B cell aplasia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with AEs and SAEs | Day 1 to 2 years
  Long term safety follow up

SECONDARY OUTCOMES:
CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Maximum observed blood concentration Cmax) | Pre-dose, up to 2 years
  Blood samples will be collected to assess cellular kinetics.
CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Area under plasma concentration -time AUC) | Pre-dose, up to 2 years
  Blood samples will be collected to assess cellular kinetics.
CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Time to reach maximum concentration Tmax) | Pre-dose, up to 2 years
  Blood samples will be collected to assess cellular kinetics.
CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Terminal elimination half-life T1/2) | Pre-dose, up to 2 years
  Blood samples will be collected to assess cellular kinetics.
CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Last measurable concentration Clast) | Pre-dose, up to 2 years
  Blood samples will be collected to assess cellular kinetics.
CAR transgene levels by quantitative polymerase chain reaction (qPCR) in blood (Time to reach last measurable concentration Tlast) | Pre-dose, up to 2 years
  Blood samples will be collected to assess cellular kinetics.
Number of patients with anti-drug antibodies | Pre-dose, up to 2 years
  Blood samples will be collected to measure anti-drug antibodies against YTB323.
Level of T cell activation by YTB323 | Pre-dose, up to 2 years
  Blood samples will be collected to measure the level of T cell activation by YTB323.
Number of patients infused with planned target dose | Day 1
  Feasibility of the manufacturing process in autoimmune disorders.
Change from pre-dose up to 2 years in the Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) score | Pre-dose, up to 2 years
  SLEDAI-2K scores are between 0 and 105, a higher score represents a higher disease activity.
Change from pre-dose up to 2 years in Physician's global assessment (PGA) | Pre-dose, up to 2 years
  The Physician's Global assessment is a visual analog scale from 0 to 3, 0 represents no activity and 3 represents severe disease activity.
Change from pre-dose up to 2 years in Lupus Low Disease Activity State (LLDAS) | Pre-dose, up to 2 years
  LLDAS is a composite measure based on: SLEDAI-2K ≤ 4, with no activity in major organ system (renal, central nervous system, cardiopulmonary, vasculitis, and fever) and no hemolytic anemia or gastrointestinal activity, current, no new lupus disease activity compared with the previous assessment, prednisone (or its equivalent) dose ≤ 7.5 mg/day, PGA (scale 0-3) ≤ 1, well tolerated standard maintenance doses of immunosuppressive lupus therapy.
Remission rate | Up to 2 years
  Remission as specified by Definitions Of Remission In Systemic Lupus Erythematosus (DORIS) criteria: Clinical SLEDAI=0, PGA<0.5 (0-3) irrespective of serology.
  The patient may be on antimalarials, low-dose glucocorticoids (prednisolone ≤5 mg/day), and/or stable immunosuppressive therapy including biologics.
Change from pre-dose up to 2 years in Urinary protein creatinine ratio (UPCR) | Pre-dose, up to 2 years
  Change in the value of UPCR.
Incidence of Complete renal response (CRR) | Up to 2 years
  Number of participants who achieved CRR.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceutical
Locations (10):
- Novartis Investigative Site, Clayton, Victoria, Australia
- France (3):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Strasbourg
- Germany (2):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Mainz
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com